CLINICAL TRIAL: NCT02731352
Title: Study of Apatinib in Patients With Local Advanced/Metastatic Iodine-131（131I）-Refractory/Resistant Differentiated Thyroid Cancer
Brief Title: Study of Apatinib in Patients With Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yansong Lin, Prof. M.D., Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-T301
Record Dates: First submitted 2016-03-07; First posted 2016-04-07 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Cancer
Keywords: apatinib; Iodine-131; Differentiated Thyroid Cancer; refractory; resistant
MeSH Terms: conditions — Thyroid Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iodine-131 Refractory/Resistant Differentiated Thyroid Cancer (Experimental): iodine-131 (131I) -Refractory/Resistant Differentiated Thyroid Cancer
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib Mesylate Tablets 750 mg q.d p.o. in 1-10 cases of differentiated thyroid cancer subjects.
  Other Names: Apatinib 750mg
Drug: Apatinib — Apatinib Mesylate Tablets 500 mg q.d. p.o. in 11-20 cases of differentiated thyroid cancer subjects.
  Other Names: Apatinib 500mg

SUMMARY:
The purpose of this study is to assess the efficacy and safety of apatinib in locally advanced/metastatic radioactive iodine-refractory/resistant differentiated thyroid cancer

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic differentiated thyroid cancer (papillary, follicular, Hurthle cells, poorly differentiated carcinoma). At least one measurable lesion (helical CT scan long diameter ≥10mm, meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST） version 1.1);
2. Disease progression within 14 months before inclusion;
3. Subjects must be 131I-refractory / resistant as defined by at least one of the following;

   * Lesions that do not demonstrate iodine uptake on any radioiodine scan
   * Subjects received a single radioactive iodine therapy within 12 months (≥ 3.7 Giga Becquerel (GBq) [≥ 100 millicurie (mCi) ]) and target lesion disease progression
   * Every two radioactive iodine treatment interval <12 months, doses ≥ 3.7 GBq [≥100 mCi], disease progress more than 12 months after at least once iodine therapy;
   * Received a total dose of radioactive iodine therapy ≥ 22.2 GBq (≥ 600 mCi)
4. main organs function is normal;
5. Eastern Cooperative Oncology Group（ECOG）Performance Status（PS） :0-2;
6. An expected survival of ≥ 3 months;
7. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug;
8. Patient has to voluntarily join the study and sign the Informed Consent Form for the study;

Exclusion Criteria:

1. Other thyroid cancer histological subtypes (such as medullary carcinoma, lymphoma or sarcoma);
2. Received VEGFR inhibitor treatment within 1 month;
3. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than ClassII; II-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class II cardiac dysfunction;
4. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
5. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 3 months;
6. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
7. Received anti-thyroid cancer chemotherapy treatment (allows the use of low-dose chemotherapy with radiation sensitizer) or thalidomide(or derivative) therapy;
8. Pregnant or lactating women;
9. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | An expected average of 8 weeks
  Disease control rate
Objective response rate (ORR) | An expected average of 8 weeks
  Objective response rate

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 43 months
  progression free survival
Overall survival (OS) | Up to approximately 48 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun D, Zhang X, Jin X, Shi C, Sun Y, Zhang Y, Liang J, Lin Y. BRAFV600E mutation is associated with better prognoses in radioactive iodine refractory thyroid cancer patients treated with multi-kinase inhibitors: a retrospective analysis of registered clinical trials. Thyroid Res. 2025 Feb 10;18(1):5. doi: 10.1186/s13044-025-00223-0. PMID 39924483
- [Derived] Lin YS, Zhang X, Wang C, Liu YQ, Guan WM, Liang J. Long-Term Results of a Phase II Trial of Apatinib for Progressive Radioiodine Refractory Differentiated Thyroid Cancer. J Clin Endocrinol Metab. 2021 Jul 13;106(8):e3027-e3036. doi: 10.1210/clinem/dgab196. PMID 33769497
- [Derived] Zhang X, Wang C, Lin Y. Pilot Dose Comparison of Apatinib in Chinese Patients With Progressive Radioiodine-Refractory Differentiated Thyroid Cancer. J Clin Endocrinol Metab. 2018 Oct 1;103(10):3640-3646. doi: 10.1210/jc.2018-00381. PMID 30053006